CLINICAL TRIAL: NCT02245269
Title: A Two-way Pharmacokinetic Interaction Study of Single-Dose Atorvastatin (LIPITOR®) With Tipranavir/Ritonavir (500mg/200mg) at Steady-State and the Effect of Antacid (MAALOX®) on the Pharmacokinetics of Single-Dose Tipranavir/Ritonavir (500mg/200mg) in Healthy Volunteers
Brief Title: Pharmacokinetics of Atorvastatin With Tipranavir/Ritonavir and the Effect of Antacid on the Pharmacokinetics of Single-Dose Tipranavir/Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.21
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Atorvastatin; aluminum hydroxide, magnesium hydroxide, drug combination

ARMS (1):
- TPV/r + Atorvastatin followed by TPV/r + antacid (Experimental): Day 1: first dose of ATV Day 8: single dose of TPV/r Day 13: single dose of TPV/r, followed by a single dose of Maalox Days 14-21: morning and evening doses of TPV/r on Day 20: second dose of ATV
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Atorvastatin; Drug: Maalox

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
Drug: Atorvastatin
Drug: Maalox — Aluminum Hydroxide; Magnesium Hydroxide; Simethicone

SUMMARY:
Study to determine the effects of combined tipranavir and ritonavir treatment (at steady-state) on the single-dose pharmacokinetics of atorvastatin, the effects of single-dose atorvastatin on the steady-state pharmacokinetics of tipranavir, and the effects of antacid on the pharmacokinetics of tipranavir

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 60 years of age inclusive
2. A Body Mass Index (BMI) between 18 and 29 kg/m2
3. Signed informed consent prior to trial participation
4. Ability to swallow numerous study medications
5. Acceptable laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity is less than or equal to Grade 1, based on the AIDS Clinical Trials Group Grading Scale
6. Acceptable medical history, physical examination and ECG, and chest X-ray (if not conducted within the last 12 months) are required prior to entering the treatment phase of the study
7. Willingness to abstain from alcohol starting 2 days prior to any administration study drug up to the end of the study. Red wine must not be ingested within 5 days prior to treatment and throughout the study
8. Willingness to abstain from the following starting 10 days prior to any administration of study drug up until the end of the study:

   • Grapefruit or grapefruit juice or products containing grapefruit juice
9. Willingness to abstain from ingesting Seville oranges, garlic supplements, St. John's Wort, or Milk Thistle, within 5 days of treatment and for the duration of the study
10. Willingness to abstain from methylxanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.) within 72 hours of each pharmacokinetic (PK) sampling day and until after the last sample from each of the intensive sampling days is collected
11. Willingness to abstain from over the counter herbal medications for the duration of the study
12. Willingness to abstain from vigorous physical exercise during PK Days
13. Reasonable probability for completion of the study

Exclusion Criteria:

1. Female subjects who are of reproductive potential who:

   * Have positive serum β-human chorionic gonadotropin at Visit 1, or on Day 0
   * Have not been using a barrier contraceptive method for at least 3 months prior to Day 0 (Visit 2)
   * Are not willing to use a reliable method of barrier contraception (such as diaphragm or condoms), during the trial and 30 days after completion/termination
   * Are breast-feeding
2. Use of any pharmacological contraceptive (including oral, patch or injectable contraceptives) for 1 month prior to study initiation and for the duration of the study
3. Use of hormone replacement therapy for 1 month prior to study initiation and for the duration of the study
4. Participation in another trial with an investigational medicine within 60 days prior to Day 0 (Visit 2)
5. Use of any medication listed in the protocol within 30 days prior to Day 0 (Visit 2)
6. Administration of antibiotics within 10 days prior to Day 0 (Visit 2) or during the trial
7. History of acute illness within the past sixty (60) days. Subjects will be excluded for these disorders greater than sixty days if, in the opinion of the investigator, the subject does not qualify as a healthy volunteer
8. Have serological evidence of Hepatitis B or C Virus
9. Have serological evidence of exposure to HIV
10. Recent history of alcohol or substance abuse (within 6 months of study period)
11. Smokers who smoke greater than 10 cigarettes or 3 cigars or 3 pipes per day; inability to refrain from smoking during the trial
12. Blood or plasma donations within 30 days prior to Day 0 (Visit 2) or during the trial
13. Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min
14. Subjects with a history of any illness or allergy that, in the opinion of the investigator,might confound the results of the study or pose additional risk in administering Tipranavir,Ritonavir, atorvastatin or erythromycin to the subject
15. Subjects who are currently taking any over-the-counter drug within 7 days prior to Day 0,(Visit 2) or who are currently taking any prescription drug that, in the opinion of the investigator in consultation with the clinical monitor, might interfere with either the absorption, distribution or metabolism of the test substances
16. Known hypersensitivity to Tipranavir,Ritonavir, sulfonamides, atorvastatin, erythromycin or saccharin
17. Inability to comply with the protocol

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2003-07; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve from time zero to infinity of the analyte (AUC0-∞) | up to day 22
Maximum plasma concentration of the analyte (Cmax) | up to day 22
Drug concentration of the analyte in plasma at 12 hours after administration (Cp12h) | up to day 22
AUC0-12 hours of the analyte | up to day 22

SECONDARY OUTCOMES:
Oral clearance (CL/F) | up to day 22
Volume of distribution (V) | up to day 22
Time of maximum concentration (tmax) | up to day 22
Apparent terminal half life (t1/2) | up to day 22
Mean Residence Time (MRT) | up to day 22
Hepatic cytochrome P450 3A4 activity using the Erythromycin Breath Test | Days 7-10
Number of patients with adverse events | up to day 22
Number of patients with clinically relevant changes in laboratory tests | up to day 22